CLINICAL TRIAL: NCT01329705
Title: Dynamic Splinting for Excessive Plantarflexion in Patients With Spastic Hemiplegia: A Randomized, Controlled Study of Gait Analysis
Brief Title: Dynamic Splinting for Plantarflexion in Spastic Hemiplegia
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Sponsor: Dynasplint Systems, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Dyna-2011
Record Dates: First submitted 2011-04-04; First posted 2011-04-06 (Estimated); Last update posted 2013-08-12 (Estimated); Status verified 2013-08

CONDITIONS: Spastic Hemiplegia
MeSH Terms: conditions — Hemiplegia | interventions — Standard of Care

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Control (Active Comparator): All patients will be treated with the current standard of care including onabotulinum toxin
  Interventions: Other: Standard of care
- Dynasplint (Experimental): Patients in the experimental Dynasplint group will be treated with the current standard of care, including onabotulinum toxin, and use the Ankle Dorsiflexion Dynasplint
  Interventions: Device: Ankle Dorsiflexion Dynasplint

INTERVENTIONS:
Device: Ankle Dorsiflexion Dynasplint — Dynamic splinting utilizes the protocols of Low-Load Prolonged Stretch (LLPS) with calibrated adjustable tension to increase Total End Range Time (TERT)to reduce contracture. The Dynasplint or "Experimental" group will add this therapy to their standard of care regimen
  Other Names: ADFD, AFD
  Arms: Dynasplint
Other: Standard of care — Patients will begin a 12 week course of physical therapy with once-weekly therapy appointment, focusing on:
  * range of motion stretching of the Achilles tendon, hamstrings, hip flexors and any other tight musculature
  * strengthening of tibialis anterior to allow dorsiflexion in swing phase of gait as well as strengthening of other weak musculature
  * gait training to improve heel strike and toe off, stride length, and gait progression
  * sensory, proprioceptive training in foot position and degree of plantarflexion or dorsiflexion
  * no electric stimulation (e-stim) will be utilized
  Arms: Control

SUMMARY:
The purpose of this study is to examine the effectiveness of onabotulinum toxin A (BTX) injections (tone management) and dynamic splinting (contracture reduction) for improving gait patterns in patients with spastic hypertnoia due to stroke or traumatic brain injury and resultant excessive plantarflexion.

ELIGIBILITY:
Inclusion Criteria:

* Patients enrolled will be male or female, be at least 18 years of age, and have been diagnosed with spastic hemiplegia and excessive plantarflexion, which includes the following:

  1. Diagnosis of a stroke or traumatic brain injury more than 6 months prior to enrollment in this study
  2. Reduced AROM and PROM in ankle dorsiflexion
  3. Ability to ambulate safely 20 feet without an ankle-foot orthosis (AFO)
  4. Inability to ambulate with initial heel-contact
  5. No prior BTX treatment within 6 months
  6. R1 of -10° or greater (using the Tardeiu method of assessment)
  7. Mean Ashworth Scale Test ≥3 for plantarflexors

Exclusion Criteria:

1. Bell's Palsy
2. Viral Encephalitis
3. Muscular Dystrophy
4. Multiple Sclerosis
5. Prior heel-cord lengthening or tendon-transfer procedure in the foot/ankle
6. Subjects with a fixed contracture of the ankle
7. Female subjects who are pregnant (positive urine pregnancy test), who have an infant they are breastfeeding, or are of childbearing potential and do not practice a reliable method of birth control
8. Bleeding disorders
9. Diagnosis of a disease that may interfere with neuromuscular function (ie. Myasthenia Gravis, Lambert-Eaton Myasthenic Syndrome, amyotrophic lateral sclerosis)
10. Subjects currently using aminoglycoside antibiotics, curare-like agents, or other agents that may interfere with neuromuscular function
11. Subjects with profound weakness or atrophy of the muscles in the target areas of injection
12. Active systemic infection or infection at the injection site
13. Allergy or sensitivity to botulinum toxin A

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2011-05; Primary Completion 2015-05 (Estimated); Study Completion 2015-08 (Estimated)

PRIMARY OUTCOMES:
Change in gait pattern | 12 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- Medical College of Wisconsin, Milwaukee, Wisconsin, United States

REFERENCES:
- [Background] Abe H, Michimata A, Sugawara K, Sugaya N, Izumi S. Improving gait stability in stroke hemiplegic patients with a plastic ankle-foot orthosis. Tohoku J Exp Med. 2009 Jul;218(3):193-9. doi: 10.1620/tjem.218.193. PMID 19561389
- [Background] Cormack J, Powers CM. Is there evidence that botulinum toxin injections are more effective than phenol injections in relieving poststroke reflex activity during plantar flexion, thereby increasing ankle range of motion and improving gait function? Phys Ther. 2004 Jan;84(1):76-84. No abstract available. PMID 14992678
- [Background] Cruz TH, Dhaher YY. Impact of ankle-foot-orthosis on frontal plane behaviors post-stroke. Gait Posture. 2009 Oct;30(3):312-6. doi: 10.1016/j.gaitpost.2009.05.018. Epub 2009 Jun 30. PMID 19570678
- [Background] Franceschini M, Carda S, Agosti M, Antenucci R, Malgrati D, Cisari C; Gruppo Italiano Studio Allevio Carico Ictus. Walking after stroke: what does treadmill training with body weight support add to overground gait training in patients early after stroke?: a single-blind, randomized, controlled trial. Stroke. 2009 Sep;40(9):3079-85. doi: 10.1161/STROKEAHA.109.555540. Epub 2009 Jun 25. PMID 19556526
- [Background] Freivogel S, Schmalohr D, Mehrholz J. Improved walking ability and reduced therapeutic stress with an electromechanical gait device. J Rehabil Med. 2009 Sep;41(9):734-9. doi: 10.2340/16501977-0422. PMID 19774307
- [Background] Johnson CA, Burridge JH, Strike PW, Wood DE, Swain ID. The effect of combined use of botulinum toxin type A and functional electric stimulation in the treatment of spastic drop foot after stroke: a preliminary investigation. Arch Phys Med Rehabil. 2004 Jun;85(6):902-9. doi: 10.1016/j.apmr.2003.08.081. PMID 15179643
- [Background] Kesar TM, Perumal R, Reisman DS, Jancosko A, Rudolph KS, Higginson JS, Binder-Macleod SA. Functional electrical stimulation of ankle plantarflexor and dorsiflexor muscles: effects on poststroke gait. Stroke. 2009 Dec;40(12):3821-7. doi: 10.1161/STROKEAHA.109.560375. Epub 2009 Oct 15. PMID 19834018
- [Background] Kim JH, Jang SH, Kim CS, Jung JH, You JH. Use of virtual reality to enhance balance and ambulation in chronic stroke: a double-blind, randomized controlled study. Am J Phys Med Rehabil. 2009 Sep;88(9):693-701. doi: 10.1097/PHM.0b013e3181b33350. PMID 19692788
- [Background] Lam T, Luttmann K, Houldin A, Chan C. Treadmill-based locomotor training with leg weights to enhance functional ambulation in people with chronic stroke: a pilot study. J Neurol Phys Ther. 2009 Sep;33(3):129-35. doi: 10.1097/NPT.0b013e3181b57de5. PMID 19809391
- [Background] Lai JM, Francisco GE, Willis FB. Dynamic splinting after treatment with botulinum toxin type-A: a randomized controlled pilot study. Adv Ther. 2009 Feb;26(2):241-8. doi: 10.1007/s12325-008-0139-2. Epub 2009 Feb 4. PMID 19194671
- [Background] John MM, Willis FB, Portillo A. Dynamic splinting for runner's toe: a case report with gait analysis. J Am Podiatr Med Assoc. 2009 Jul-Aug;99(4):367-70. doi: 10.7547/0980367. PMID 19605933
- [Background] Masiero S, Briani C, Marchese-Ragona R, Giacometti P, Costantini M, Zaninotto G. Successful treatment of long-standing post-stroke dysphagia with botulinum toxin and rehabilitation. J Rehabil Med. 2006 May;38(3):201-3. doi: 10.1080/16501970500515840. PMID 16702088
- [Background] McGuire JR. Effective use of chemodenervation and chemical neurolysis in the management of poststroke spasticity. Top Stroke Rehabil. 2001 Spring;8(1):47-55. doi: 10.1310/CYP4-BPXC-CG8M-XCA3. PMID 14523751
- [Background] Michael K, Goldberg AP, Treuth MS, Beans J, Normandt P, Macko RF. Progressive adaptive physical activity in stroke improves balance, gait, and fitness: preliminary results. Top Stroke Rehabil. 2009 Mar-Apr;16(2):133-9. doi: 10.1310/tsr1602-133. PMID 19581199
- [Background] Pleis JR, Lucas JW, Ward BW. Summary health statistics for U.S. adults: National Health Interview Survey, 2008. Vital Health Stat 10. 2009 Dec;(242):1-157. PMID 20821903
- [Background] States RA, Pappas E, Salem Y. Overground physical therapy gait training for chronic stroke patients with mobility deficits. Cochrane Database Syst Rev. 2009 Jul 8;2009(3):CD006075. doi: 10.1002/14651858.CD006075.pub2. PMID 19588381
- [Background] Stock R, Mork PJ. The effect of an intensive exercise programme on leg function in chronic stroke patients: a pilot study with one-year follow-up. Clin Rehabil. 2009 Sep;23(9):790-9. doi: 10.1177/0269215509335291. Epub 2009 Jun 26. PMID 19561034
- [Background] Usuba M, Akai M, Shirasaki Y, Miyakawa S. Experimental joint contracture correction with low torque--long duration repeated stretching. Clin Orthop Relat Res. 2007 Mar;456:70-8. doi: 10.1097/BLO.0b013e31803212bf. PMID 17224840
- [Background] Willis, F. B. Post-TBI Gait Rehabilitation. Applied Neurol. 2007 Jul;3(7):25-26.
- [Background] Lai JM, Jones M, and Willis FB. Effect of Dynamic Splinting on Excessive Plantarflexion Tone/Contracture: A Controlled, Crossover Study. Proceedings of the 16th European Congress of Physical and Rehabilitation Medicine. Minerva Medica pubs, Italy, August 2008, pg 106-109.
- [Background] Miller EL, Murray L, Richards L, Zorowitz RD, Bakas T, Clark P, Billinger SA; American Heart Association Council on Cardiovascular Nursing and the Stroke Council. Comprehensive overview of nursing and interdisciplinary rehabilitation care of the stroke patient: a scientific statement from the American Heart Association. Stroke. 2010 Oct;41(10):2402-48. doi: 10.1161/STR.0b013e3181e7512b. Epub 2010 Sep 2. No abstract available. PMID 20813995
- [Background] Lloyd-Jones D, Adams R, Carnethon M, De Simone G, Ferguson TB, Flegal K, Ford E, Furie K, Go A, Greenlund K, Haase N, Hailpern S, Ho M, Howard V, Kissela B, Kittner S, Lackland D, Lisabeth L, Marelli A, McDermott M, Meigs J, Mozaffarian D, Nichol G, O'Donnell C, Roger V, Rosamond W, Sacco R, Sorlie P, Stafford R, Steinberger J, Thom T, Wasserthiel-Smoller S, Wong N, Wylie-Rosett J, Hong Y; American Heart Association Statistics Committee and Stroke Statistics Subcommittee. Heart disease and stroke statistics--2009 update: a report from the American Heart Association Statistics Committee and Stroke Statistics Subcommittee. Circulation. 2009 Jan 27;119(3):480-6. doi: 10.1161/CIRCULATIONAHA.108.191259. No abstract available. PMID 19171871
- [Background] Sheean G. Neurophysiology of spasticity. In: Barnes MP, Johnson GR. Upper motor neuron syndrome and spasticity. Cambridge University Press, 2008: 9-63.
- [Background] Hesse S, Lucke D, Malezic M, Bertelt C, Friedrich H, Gregoric M, Mauritz KH. Botulinum toxin treatment for lower limb extensor spasticity in chronic hemiparetic patients. J Neurol Neurosurg Psychiatry. 1994 Nov;57(11):1321-4. doi: 10.1136/jnnp.57.11.1321. PMID 7964805
- [Background] Pittock SJ, Moore AP, Hardiman O, Ehler E, Kovac M, Bojakowski J, Al Khawaja I, Brozman M, Kanovsky P, Skorometz A, Slawek J, Reichel G, Stenner A, Timerbaeva S, Stelmasiak Z, Zifko UA, Bhakta B, Coxon E. A double-blind randomised placebo-controlled evaluation of three doses of botulinum toxin type A (Dysport) in the treatment of spastic equinovarus deformity after stroke. Cerebrovasc Dis. 2003;15(4):289-300. doi: 10.1159/000069495. PMID 12686794
- [Background] Harvey L, Herbert R, Crosbie J. Does stretching induce lasting increases in joint ROM? A systematic review. Physiother Res Int. 2002;7(1):1-13. doi: 10.1002/pri.236. PMID 11992980